CLINICAL TRIAL: NCT05186636
Title: Dialyzing Wisely - Improving the Delivery of Acute Renal Replacement Therapy to Albertans
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00112499
Record Dates: First submitted 2021-12-09; First posted 2022-01-11 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Acute Renal Injury
Keywords: evidence based care pathway,; critical care medicine; quality improvement; acute renal replacement therapy
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients receiving renal replacement therapy: All patients in participating ICU's receiving CRRT or IRRT during the study period
  Interventions: Other: KPI reports; Other: Prescriber reports

INTERVENTIONS:
Other: KPI reports — Quarterly
  Other Names: Monitoring, reporting and regular review of acute RRT KPIs
Other: Prescriber reports — Individualized prescriber reports for acute RRT initiation patterns along with targeted education to ensure that align with best evidence-based practices

SUMMARY:
Implementation of an evidence-based and best practices acute RRT pathway aiming to decrease acute RRT program and healthcare systems costs while improving important patient-reported outcomes.

DETAILED DESCRIPTION:
Providing acute dialysis to critically ill patients in ICU settings is resource and cost intensive. The daily costs of acute dialysis can range from $528/day for intermittent hemodialysis to $865/day for continuous renal replacement therapy. Providing acute dialysis in ICU settings requires a specialized team of nurses, educators, physicians and stakeholders to ensure its safe and effective prescription and delivery. Acute dialysis is typically delivered to some of the most acutely ill patients admitted to the ICU to support organ function and sustain life.

At present, there is not a standardized approach to the prescription and delivery of acute dialysis therapy in ICUs across Alberta. The DIALYZING WISELY program will implement a standardized approach to the delivery of best practices for acute dialysis therapy to all patients who receive treatment across ICUs in Alberta.

ELIGIBILITY:
Inclusion Criteria:

Patient in one of 15 adult and 3 pediatric intensive care units in Alberta Receive acute RRT as part of their usual clinical care during the intervention period

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients from 15 adult and 3 pediatric Alberta ICUs who receive acute RRT as part of their usual clinical care during the intervention period
Sampling Method: Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Key performance indicators (KPI) | Throughout intervention period up to 3 years
  Changes in acute KPIs
Health system costs | 3 years
  Acute RRT and healthcare systems costs

SECONDARY OUTCOMES:
Length of renal replacement therapy | 3 years
  Length of time patient receives RRT during their ICU stay
ICU and hospital lengths of stay | 3 years
  Number of days patient spends in the ICU and hospital
ICU and 90 day mortality | 3 years
  number of patients who die before ICU discharge or within 90 days of ICU stay
Rates of RRT dependence at 90 days | 3 years
  number of patients who are receiving RRT at 90 days after ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Oleksa Rewa, MD, Principal Investigator — University of Alberta
Locations (15):
- Canada (15):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - Alberta Children's Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Manzankowski Alberta Heart Institute, Edmonton, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Grande Prairie Regional Hospital, Grande Prairie, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Red Deer Regional Hospital Centre, Red Deer, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta

REFERENCES:
- [Derived] Opgenorth D, Bagshaw SM, Lau V, Graham MM, Fraser N, Klarenbach S, Morrin L, Norris C, Pannu N, Sinnadurai S, Valaire S, Wang X, Rewa OG. A study protocol for improving the delivery of acute kidney replacement therapy (KRT) to critically ill patients in Alberta - DIALYZING WISELY. BMC Nephrol. 2022 Nov 16;23(1):369. doi: 10.1186/s12882-022-02990-6. PMID 36384465